CLINICAL TRIAL: NCT02216890
Title: A Phase 1 Trial of SGN-CD70A in Patients With CD70-Positive Malignancies
Brief Title: Safety Study of SGN-CD70A in Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGN70A-001
Record Dates: First submitted 2014-08-12; First posted 2014-08-15 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Renal Cell Carcinoma; Mantle-Cell Lymphoma; Diffuse, Large B-Cell, Lymphoma; Follicular Lymphoma, Grade 3
Keywords: Renal Cell Carcinoma; Mantle-Cell Lymphoma; Diffuse, Large B-Cell, Lymphoma; Follicular Lymphoma, Grade 3; Antibody-Drug Conjugate; CD70 Antigen; Drug Therapy
MeSH Terms: conditions — Carcinoma, Renal Cell; Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SGN-CD70A (Experimental)
  Interventions: Drug: SGN-CD70A

INTERVENTIONS:
Drug: SGN-CD70A — Given intravenously every 3 weeks (or an alternate dosing schedule up to every 6 weeks)

SUMMARY:
This study will examine the safety profile of SGN-CD70A. The study will test increasing doses of SGN-CD70A given every 3 weeks (or an alternate dosing schedule up to every 6 weeks) to small groups of patients. The goal is to find the highest dose of SGN-CD70A that can be given to patients without causing unacceptable side effects. The pharmacokinetics and antitumor activity of SGN-CD70A will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic renal cell carcinoma, mantle cell lymphoma, or diffuse large B-cell lymphoma including Grade 3b follicular lymphoma
* Relapsed, refractory, or progressive disease following at least 2 prior systemic therapies
* Confirmed positive CD70 expression on tumor tissue
* Eastern Cooperative Oncology Group performance status 0 or 1
* Adequate baseline hematologic, pulmonary, renal, and hepatic function
* Measurable disease

Exclusion Criteria:

* Prior treatment with anti-CD70 directed therapy unless CD70 expression is confirmed on tumor tissue obtained after the treatment
* Patients <100 days since prior allogeneic stem cell transplant
* Less than 4 weeks since prior treatment; or 2 weeks if patient experienced disease progression on the prior treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2017-02-15 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Through 1 month following last dose
Incidence of laboratory abnormalities | Through 1 month following last dose

SECONDARY OUTCOMES:
Blood concentrations of SGN-CD70A and metabolites | Through 3 to 6 weeks after dosing
Incidence of antitherapeutic antibodies | Through 1 month following last dose
Objective response rate | Through 1 month following last dose
Progression-free survival | Approximately 3 years
Duration of response | Approximately 3 years

OTHER OUTCOMES:
Exploratory biomarkers of pharmacodynamic effects due to SGN-CD70A | Through 1 month following last dose

CONTACTS AND LOCATIONS:
Overall Officials: Elaina Gartner, MD, Study Director — Seagen Inc.
Locations (17):
- United States (17):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - Cardinal Bernardin Cancer Center / Loyola University Medical Center, Maywood, Illinois
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Karmanos Cancer Institute / Wayne State University, Detroit, Michigan
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - James P. Wilmot Cancer Center / University of Rochester Medical Center, Rochester, New York
  - UNC Lineberger Comprehensive Cancer Center / University of North Carolina, Chapel Hill, North Carolina
  - University of Cincinnati Cancer Institute, Cincinnati, Ohio
  - Case Western Reserve University / University Hospitals Case Medical Center, Cleveland, Ohio
  - University of Pennsylvania / Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Medical University of South Carolina/Hollings Cancer Center, Charleston, South Carolina
  - Texas Oncology - Austin Midtown, Austin, Texas
  - Methodist Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Seattle Cancer Care Alliance / University of Washington, Seattle, Washington
  - Northwest Cancer Specialists, P.C., Vancouver, Washington